CLINICAL TRIAL: NCT06115252
Title: Partnering to Enhance Emerging Adults' Response to Programs (PEER)
Brief Title: Partnering to Enhance Emerging Adults' Response to Programs
Acronym: PEER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: University of Texas (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sarah Feldstein Ewing, Professor, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: O25-013-1; 1R01AA030678-01 (NIH)
Record Dates: First submitted 2023-10-17; First posted 2023-11-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use, Unspecified
MeSH Terms: conditions — Alcohol Drinking | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Motivational Interviewing (MI) (Experimental)
  Interventions: Behavioral: Motivational Interviewing (MI)

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — Motivational interviewing with peer dyads starts with an open-ended exploration of the dyad's hazardous drinking behavior via personal stories about alcohol use. It includes a values clarification task and age-matched norms along with personalized feedback regarding the dyad's alcohol use. The goal of the session is to engage the dyad in a thoughtful conversation about drinking and the implications it may have on their lives, with an eye to bolstering and supporting inherent drive for behavior change.

SUMMARY:
The goal of this clinical trial (CT) is to learn more about emerging adults' and their peers. Here, we will see how co-participating with a peer in health program might impact brain and behavior change over time.

Eligible youth will be invited to come in for a "Participation Day," during which they and a peer will independently complete questionnaires. With a peer, they will then complete a short health program, and undergo a brain scan (fMRI) while completing activities. Our study team will reach out to each participant individually again 3, 6, and 12 months later to learn about health behaviors over time.

ELIGIBILITY:
Inclusion Criteria:

* within the specified age range
* agree to be contacted for the 3, 6, and 12 month follow ups
* provide fully informed consent

Exclusion Criteria:

* left-handed
* evidence of brain injury/illness and/or neurological, neurodevelopmental disorder including psychosis and related medications (e.g., antipsychotics; neuroleptics)
* loss of consciousness ≥ 2 minutes
* other fMRI contraindications (e.g., unremovable metal on/in body, pregnant)

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 248 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Blood oxygen level dependent (BOLD) response synchrony | Baseline
  Mean BOLD time series will be obtained for each region of interest (ROI) during peer-directed change talk trials and temporally aligned across dyad participants. Inter-brain synchrony will be quantified using z-transformed GLM β-weights within ROIs between the BOLD time series of dyad members.
BOLD response synchrony association with behavior change (past month alcohol use days) | 12 Months
  Pearson correlation coefficients (r) of Primary Outcome #1 (ROI z-scores representing BOLD response synchrony) with individual Timeline Followback (TLFB) past month drinking days at 12 month follow up.

SECONDARY OUTCOMES:
BOLD response synchrony association with behavior change (past month alcohol use days) | 3 Months
  Pearson correlation coefficients (r) of Primary Outcome #1 (ROI z-scores representing BOLD response synchrony) with individual Timeline Followback (TLFB) past month drinking days at 3 month follow up.
BOLD response synchrony association with behavior change (past month alcohol use days) | 6 Months
  Pearson correlation coefficients (r) of Primary Outcome #1 (ROI z-scores representing BOLD response synchrony) with individual Timeline Followback (TLFB) past month drinking days at 6 month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah W. Feldstein Ewing, PhD, Principal Investigator — UConn Health; Francesca Filbey, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will submit and share data with the NIAAA Data Archive, a data repository housed within the NIMH Data Archive, and will follow the guidelines described in NOT-AA-23-002.
Supporting Information: Study Protocol
Time Frame: Data will be submitted on or before the NDA submission due dates and maintained for the duration required by NIAAA Data Archive Data Sharing Plan.
Access Criteria: See details provided by the NIAAA Data Archive.
URL: https://nda.nih.gov/niaaa